CLINICAL TRIAL: NCT00361842
Title: Multicenter, Open-Label, Phase 2 Study Of CPX-1 (Irinotecan HCl: Floxuridine) Liposome Injection In Patients With Advanced Colorectal Carcinoma
Brief Title: Multicenter Study Of CPX-1 (Irinotecan HCl: Floxuridine) Liposome Injection In Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol CLTR0105-201
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal cancer; Colorectal carcinoma; Colonic cancer; Rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Liposomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan (Experimental)
  Interventions: Drug: CPX-1 (Irinotecan HCl:Floxuridine) Liposome Injection

INTERVENTIONS:
Drug: CPX-1 (Irinotecan HCl:Floxuridine) Liposome Injection — CPX-1 Liposome Injection is a liposomal formulation of a fixed combination of the antineoplastic drugs irinotecan HCl and floxuridine.

SUMMARY:
The purpose of this study is to determine whether CPX-1 is effective in patients with advanced colorectal cancer who have already received chemotherapy that included the drug oxaliplatin or irinotecan. All patients will receive CPX-1 at a dose of 210 units/m2 over 90 minutes every two weeks.

DETAILED DESCRIPTION:
CPX-1 Liposome Injection is a liposomal formulation of a fixed combination of the antineoplastic drugs irinotecan HCl and floxuridine. The two drugs are present inside the liposome in a fixed 1:1 molar ratio. CPX-1 was developed as a means of delivering and preserving a fixed 1:1 molar ratio of the two drugs. This ratio was found in vitro and in vivo models of cancer to have synergistic anti-cancer activity and preservation and delivery of this ratio is important because other ratios of these two drugs have been found to be antagonistic or only additive. Both floxuridine and irinotecan HCl are active chemotherapeutic agents, each approved for clinical use in the United States and Canada for colorectal cancer. Current practice routinely administers 5- fluorouracil with irinotecan in combination regimens in first or second line treatment without the means of preserving the synergistic ratio.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily sign an informed consent form
* Age > 18 years at the time of signing the informed consent form
* Histological confirmation of advanced stage, primary or metastatic colorectal carcinoma
* Prior therapy (Group 1, irinotecan naive):

  * No more than one regimen for metastatic disease
  * No more than two regimens overall; one for neoadjuvant/adjuvant and one for metastatic/advanced disease
* Prior therapy (Group 2, irinotecan refractory):

  * Disease progression on or within 3 months after prior irinotecan-containing regimen
  * CPX-1 treatment must start within 6 months after documentation of disease progression on irinotecan (other therapies are permitted after irinotecan and before study entry)
* Must have measurable disease as defined by RECIST
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Able to adhere to the study visit schedule and other protocol requirements
* Life expectancy of at least 24 weeks
* Laboratory values fulfilling the following:

  * Absolute neutrophil count (ANC) >1500 cells/mm3 (1.5 x 109/L)
  * Platelet count > 100,000/mm3 (100 x 109/L)
  * Serum creatinine <1.5 x upper limits of normal (ULN)
  * Serum SGOT/AST and SGPT/ALT <3 x upper limits of normal (ULN) (<5 times ULN if caused by liver metastases)
  * Serum total bilirubin < 1.25 x upper limits of normal (<2 times ULN if caused by liver metastases)
* All men and women must agree to practice effective contraception during the study period and for three months afterward if not otherwise documented to be infertile.
* Prior radiation therapy must be completed at least 4 weeks prior to enrollment and the patient recovered from any toxicity related to the radiation therapy.

Exclusion Criteria:

* Prior treatment with irinotecan or an irinotecan-containing regimen (Group 1 only)
* Intolerant of an irinotecan-containing regimen (Group 2 only)
* Without documented evidence of irinotecan-refractoriness (Group 2 only)
* Chemotherapy or investigational anticancer therapeutic drugs in the four weeks prior to study entry.
* Hypersensitivity to irinotecan, floxuridine or liposomal products.
* History of Wilson's disease or other copper-related disorder.
* Clinically significant cardiac disease (New York Heart Association Class III or IV).
* Severe debilitating pulmonary disease.
* Active infection requiring continuing intravenous antibiotic treatment; recent infections must have resolved at least 5 days
* Severe or active enteropathy or recurrent onset of diarrhea, defined as an excess of 2 to 3 stools above the normal daily rate within the past four weeks.
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating women. Continued use of a drug or other product known to induce or inhibit CYP3A4. ---Patients must discontinue these products for at least 2 week prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital; John Marshall, MD, Principal Investigator — Lombardi Comprehensive Cancer Center, Georgetown University Medical Center; Arthur Louie, MD, Study Director — Jazz Pharmaceuticals
Locations (13):
- United States (11):
  - California Cancer Center, Greenbrae, California
  - Lombardi Comprehensive Cancer Research Institute, Georgetown University Medical Center, Washington D.C., District of Columbia
  - NW Oncology & Hematology Associates, Coral Springs, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - St. Joseph's/Candler Health System Inc., Savannah, Georgia
  - Presbyterian Hospital, Charlotte, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Cancer Care Oklahoma, Oklahoma City, Oklahoma
  - Cancer Care Oklahoma, Tulsa, Oklahoma
  - South Carolina Oncology Association, Columbia, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Irinotecan - Naïve | Irinotecan - Exposed
Started | 28 | 35
Completed | 1 | 1
Not Completed | 27 | 34
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 2 | 1
Not completed — Disease progression | 19 | 20
Not completed — Adverse Event | 2 | 3
Not completed — Occurrence of unacceptable toxicity | 1 | 5
Not completed — Other | 1 | 0
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled participants who received at least one dose of CPX 1. The total number of participants in the safety analysis set was 59 (26 in group 1, irinotecan-naïve and 33 in group 2, irinotecan-exposed).
Groups:
- Total: Total of all reporting groups
Arm/Group | Irinotecan - Naïve | Irinotecan - Exposed | Total
Number analyzed (Participants) | 26 | 33 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.62) | 60.2 (10.92) | 60.1 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 13 | 18 | 31
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 17 | 25
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0
Description: Disease response was assessed using RECIST 1.0. Measurable disease and target lesions were determined prior to study entry. Changes in the largest diameter (unidimensional measurement) of the sum of the target tumor lesions were used in the RECIST criteria. Best response on study was classified as follows. Complete Response (CR), disappearance of all clinical and radiological evidence of tumor. Partial Response (PR) at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum of the longest diameters. Stable Disease (SD), steady state of disease. Neither sufficient shrinkage to qualify for PR or sufficient increase to qualify for PD. Progressive Disease (PD) at least a 20% increase in the sum of the longest diameters of measured lesions taking as references the smallest sum of longest diameters recorded since the treatment started. Appearance of new lesions also constituted progressive disease.
Time Frame: From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
Population: The response rate efficacy evaluable (RECIST) analysis set (n=21 in group 1 and n= 24 in group 2) included all enrolled participants who received at least 1 cycle of CPX-1 therapy (2 doses, Days 1 and 15) and had at least 1 measurable lesion assessed for response (either after every second cycle of treatment or earlier to document disease progression) after beginning treatment. Tumor response, based on the RECIST criteria, was assessed at baseline and every 8 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Irinotecan - Naïve: * No prior exposure to irinotecan
  * No more than 1 regimen for metastatic disease
  * No more than 2 regimens overall;
  * 1 for neoadjuvant/adjuvant and 1 for metastatic/advanced disease
- Irinotecan - Exposed: * Prior exposure to irinotecan was required
  * Disease progression on or within 6 months after completion of prior irinotecan-containing regimen
  * CPX-1 treatment must start within 12 months after documentation of disease progression on irinotecan (other therapies are permitted after irinotecan and before study entry)
Arm/Group | Irinotecan - Naïve | Irinotecan - Exposed
Number analyzed (Participants) | 21 | 24
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 2 | 0
  Stable Disease (SD) | 11 | 12
  Progressive Disease (PD) | 8 | 11

2. Primary Outcome: Progression-free Survival (PFS) Per RECIST Version 1.0
Description: Progression-free survival (PFS) was defined as the time from the first dose to the documentation of progressive disease (PD), death, or lost to follow-up at last assessment visit.
Time Frame: Every 8 weeks
Population: The efficacy evaluable analysis set or "Full Analysis Set" (25 patients in Group 1 and 32 participants in Group 2) included all enrolled participants who received at least 1 dose of CPX-1 therapy, and had at least one post-baseline PFS assessment.
Measure: Mean (Standard Error); unit: months
Arm/Group | Irinotecan - Naïve | Irinotecan - Exposed
Number analyzed (Participants) | 25 | 32
months | 4.69 (0.84) | 3.48 (0.44)

3. Secondary Outcome: Duration of Response (DoR) Per RECIST Version 1.0
Description: The duration of overall response was measured from the time that measurement criteria were met for CR or PR (whichever status was recorded first) until the first date that recurrent or progressive disease was objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The duration of overall complete response was measured from the time measurement criteria were first met for complete response until the first date that recurrent disease was objectively documented.
Time Frame: Every 8 weeks
Population: No participants had CR. Two participants in the naïve group had objective responses. One participant showed a PR on study day 57 that lasted for 5.8 months. One participant had a PR starting on study day 60 and persisting for 9.1 months at which time the data was censored. Due to the censored observation, the median DoR was not estimable (NE).
Measure: Median (Full Range); unit: months
Arm/Group | Irinotecan - Naïve | Irinotecan - Exposed
Number analyzed (Participants) | 2 | 0
months | NA [5.8 to 9.1] — One participant had a PR starting on study day 60 and persisting for 9.1 months at which time the data was censored. Due to the censored observation, the median DoR was not estimable (NE). |

ADVERSE EVENTS:
Arm/Group | Irinotecan - Naïve | Irinotecan - Exposed
All-Cause Mortality (participants affected / at risk) | 2/26 | 4/33
Serious Adverse Events (participants affected / at risk) | 13/26 | 11/33
Other Adverse Events (participants affected / at risk) | 26/26 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan - Naïve (N=26) | Irinotecan - Exposed (N=33)
Diarrhea (Gastrointestinal disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Pyrexia (Gastrointestinal disorders) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Cardio-respiratory Arrest (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
GI Hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Small Intestine Obstruction (Gastrointestinal disorders) | 0 | 1
General Physical Deterioration (General disorders) | 1 | 0
Infusion Related Reaction (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1
GI Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1
Metastasis to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Disease Progression (General disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Irinotecan - Naïve (N=26) | Irinotecan - Exposed (N=33)
Anemia (Blood and lymphatic system disorders) | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 5 | 14
Abdominal Pain (Gastrointestinal disorders) | 10 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 7 | 8
Diarrhea (Gastrointestinal disorders) | 22 | 26
Dry Mouth (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Flatulence (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 21 | 24
Vomiting (Gastrointestinal disorders) | 18 | 17
Asthenia (General disorders) | 6 | 3
Chills (General disorders) | 4 | 3
Fatigue (General disorders) | 15 | 22
Mucosal Inflammation (General disorders) | 2 | 3
Edema, Peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 4 | 8
Nasopharyngitis (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 3
Neutrophil Count Decreased (Investigations) | 0 | 3
Weight Decreased (Investigations) | 6 | 11
Anorexia (Metabolism and nutrition disorders) | 10 | 13
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 8 | 6
Hypokalemia (Metabolism and nutrition disorders) | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 5 | 6
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnea, Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 5
Hot Flush (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.